CLINICAL TRIAL: NCT05661981
Title: A Post Market Multicenter Clinical Investigation of GLYCAR Bovine Pericardial Patch With EnCap™ Technology in Cardiac and Vascular Repair or Reconstruction Surgery. GLYCAR Study
Brief Title: GLYCAR Post Market Multicenter Study
Acronym: CIP002
Status: Active, not recruiting | Type: Observational
Sponsor: GLYCAR SA (Pty) Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: GLYCAR
Record Dates: First submitted 2022-12-07; First posted 2022-12-22 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Congenital Premature Cardiac Closure; Cardiac and Great Vessel Reconstruction and Repair; Peripheral Vascular Reconstruction and Repair
Keywords: Bovine pericardial patch

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Adult and pediatric patients: Undergoing cardiac and/or vascular repair or reconstruction surgery
  Interventions: Device: GLYCAR Pericardial Patch

INTERVENTIONS:
Device: GLYCAR Pericardial Patch — The Glycar patches are intended to be used by surgeons specialized in the field of cardiovascular surgery. The patch is intended to be used for pericardial closure, or repair and/or reconstruction of cardiovascular structures by replacing missing tissue, reinforcing weakened tissue and providing extra strength to repair tissue during healing.

SUMMARY:
Prospective, non-interventional, observational, multi-center, single arm, post market clinical follow-up study

DETAILED DESCRIPTION:
This real-world, single-arm, multi-center, observational, non-interventional prospective registry will enroll up to 100 consecutive subjects undergoing cardiac and/or vascular repair or reconstruction surgery in 10-12 investigative sites in the European Union (EU), South Africa and USA. The study is aimed at providing real-world evidence of the Glycar Pericardial patch device performance and incidence of clinical outcomes in patients undergoing cardiac and/or vascular repair or reconstruction surgery related to Glycar Pericardial patch.

ELIGIBILITY:
Inclusion Criteria:

* Patients (to be) treated with Glycar Pericardial patch as per IFU and standard clinical practice.
* The patient or patient's legal representative signs an EC/ IRB approved informed consent form prior to the study participation

Intraprocedural inclusion:

GLYCAR Pericardial Patch was implanted, or implantation attempted during the index procedure.

Exclusion Criteria:

* No study specific exclusion criteria: patients treated per standard clinical practice and do not present any of the contraindications detailed in the IFU.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This real-world, single-arm, multi-center, observational, non-interventional prospective registry will enrol up to a total of 100 consecutive subjects undergoing cardiac and/or vascular repair or reconstruction surgery in 10-12 investigative sites in the European Union (EU), South Africa and USA. The study is aimed at providing real-world evidence of the Glycar Pericardial patch device performance and incidence of clinical outcomes in patients undergoing cardiac and/or vascular repair or reconstruction surgery related to Glycar Pericardial patch.
Sampling Method: Probability Sample
Enrollment: 110 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2026-06 (Estimated); Study Completion 2027-06 (Estimated)

PRIMARY OUTCOMES:
Incidence of Glycar- Pericardial patch related mortality | 30 days post procedure or hospital discharge (whichever comes first)
  Patch related mortality at acute follow up will be determined
Incidence of Glycar- Pericardial patch related reintervention | 30 days post procedure or hospital discharge (whichever comes first)
  Patch related re-intervention at acute follow up will be determined

SECONDARY OUTCOMES:
Incidence of Glycar Pericardial patch related mortality | 1- and 2-years post-procedure
  Patch related mortality at long term follow up will be determined
Incidence of Glycar Pericardial patch related reinterventions | 1- and 2-years post-procedure
  Patch related reintervetion at long term follow up will be determined
Total number of unplanned reoperations required in patients | 30 days post procedure or hospital discharge (whichever comes first), 1- and 2-years post-procedure
  The total number of unplanned reoperations required in patients over the FU period which include the repair or alteration of the surgical area around the patch. (Patients with planned reoperations at the time of the primary index procedure will not be considered)
Incidence of thrombus formation | 30 days or hospital discharge (whichever comes first) and 1- and 2- year follow-up
  Number of thrombus formed post procedure will be taken in to account
Incidence of Glycar Pericardial Patch related unanticipated adverse events | 30 days or hospital discharge (whichever comes first) and 1- and 2-years follow-up
  Incidence rate of unanticipated adverse events reported for this patch during the FU period will be reported
Rate of detected Patch infection (such as endocarditis) | 30 days or hospital discharge (whichever comes first) and 1- and 2- year follow-up
  Any patch related infection rate will be analyzed

CONTACTS AND LOCATIONS:
Overall Officials: Julien Guihaire, Principal Investigator — Cardiac Surgeon, Head of Heart Transplantation and Mechanical Circulatory Support Program
Locations (4):
- Marie Lannelongue Hospital, Le Plessis-Robinson, France
- Germany (3):
  - Leipzig Heart Institute GmbH, Leipzig
  - German Heart Center Munich (Deutsches Herzzentrum München)- Adult Section, Munich
  - German Heart Center Munich (Deutsches Herzzentrum München)- Pediatric Section, Munich

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Bedard DL, Unterman R, Bopp LH, Brennan MJ, Haberl ML, Johnson C. Rapid assay for screening and characterizing microorganisms for the ability to degrade polychlorinated biphenyls. Appl Environ Microbiol. 1986 Apr;51(4):761-8. doi: 10.1128/aem.51.4.761-768.1986. PMID 3085588
- [Background] Hackam DJ, Rotstein OD. Stoma closure and wound infection: an evaluation of risk factors. Can J Surg. 1995 Apr;38(2):144-8. PMID 7728668
- [Background] Featherstone HJ. Headaches and heart disease: the lack of a positive association. Headache. 1986 Jan;26(1):39-41. doi: 10.1111/j.1526-4610.1986.hed2601039.x. No abstract available. PMID 3781826
- [Background] Okada N, Wada K, Goldsmith BA, Koizumi S. SHP-2 is involved in neurotrophin signaling. Biochem Biophys Res Commun. 1996 Dec 13;229(2):607-11. doi: 10.1006/bbrc.1996.1851. PMID 8954945
- [Background] Figdor PP, Todoroff K, Wiltschke H. [Acute renal failure in dysglobulinemias (multiple myeloma and amyloidosis)]. Urol Int. 1967;22(5):390-8. doi: 10.1159/000279503. No abstract available. German. PMID 6081367
- [Background] Tsai JW, Ayubi FS, Rice RD, Zhang Z, Armstrong PJ. Permacol (porcine dermal collagen) and Alloderm (acellular cadaveric dermis) as a vascular patch repair for common carotid arteriotomy in a rabbit model. Ann Vasc Surg. 2009 May-Jun;23(3):374-81. doi: 10.1016/j.avsg.2008.10.004. Epub 2008 Dec 6. PMID 19059755
- [Background] Chlupac J, Filova E, Bacakova L. Blood vessel replacement: 50 years of development and tissue engineering paradigms in vascular surgery. Physiol Res. 2009;58 Suppl 2:S119-S140. doi: 10.33549/physiolres.931918. PMID 20131930
- [Background] Edenfield L, Blazick E, Eldrup-Jorgensen J, Healey C, Bloch P, Hawkins R, Aranson N, Nolan B. Outcomes of carotid endarterectomy in the Vascular Quality Initiative based on patch type. J Vasc Surg. 2020 Apr;71(4):1260-1267. doi: 10.1016/j.jvs.2019.05.063. Epub 2019 Sep 3. PMID 31492613
- [Background] Burla L, Schwegler I, Weibel P, Weber M, Zientara A, Attigah N. Intraoperatively self-made bovine pericardial graft for portomesenteric reconstruction in pancreatic surgery. Langenbecks Arch Surg. 2020 Aug;405(5):705-712. doi: 10.1007/s00423-020-01920-0. Epub 2020 Jun 30. PMID 32607839